CLINICAL TRIAL: NCT01033214
Title: A Phase I Feasibility Study of the TAArget Thoracic Stent Graft for the Treatment of Aneurysms in the Descending Thoracic Aorta
Brief Title: ENTRUST - TAArget® Thoracic Stent Graft Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Duke Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMV-TAA-P1-001
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: TAA; Thoracic; Descending Thoracic Aorta; TAArget
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAArget Thoracic Stent Graft (Experimental): those treated with the investigational device
  Interventions: Device: Endovascular repair of TAA in the descending Thoracic Aorta

INTERVENTIONS:
Device: Endovascular repair of TAA in the descending Thoracic Aorta — Usage of the TAArget thoracic stent graft for treatment of TAA in the Descending Thoracic Aorta.

SUMMARY:
Evaluate the safety and effectiveness of endovascular repair with the LeMaitre TAArget thoracic stent graft as an alternative to open surgical repair.

DETAILED DESCRIPTION:
* Subject is > 18 years of age.
* Females subjects must be either documented post-menopausal, surgically incapable of bearing children, or for women of childbearing potential, using barrier contraceptive methods and must have a negative serum pregnancy test at screening.
* Subject is a candidate for endovascular thoracic aortic repair.
* Subject has a TAA that meets one of the following criteria:
* Is diagnosed with a Fusiform Focal TAA >5cm, or
* Is diagnosed with a Fusiform Focal TAA that has a diameter < 5 cm and has exhibited rapid expansion, or
* Is diagnosed with a Fusiform Focal TAA that has a diameter ≥ 4.5 cm and is at least twice the size of the normal DTA, or
* Is diagnosed with a saccular TAA of any size.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age. Female subjects are either documented post-menopausal, surgically incapable of bearing children, or for women of childbearing potential, using barrier contraceptive methods and have a negative serum pregnancy test at screening.

Subject is a candidate for endovascular thoracic aortic repair.

Subject has a TAA that meets one of the following criteria:

1. Is diagnosed with a Fusiform Focal TAA ≥5cm, or
2. Is diagnosed with a Fusiform Focal TAA that has a diameter ≤ 5 cm and has exhibited rapid expansion, or
3. Is diagnosed with a Fusiform Focal TAA that has a diameter ≥ 4.5 cm and is at least twice the size of the normal DTA, or
4. Is diagnosed with a saccular TAA of any size (where potential for rupture is increased*).

   * Tortuosity and angulation do not exceed 90 degrees.
   * Subject has an arterial access site that allows for the introduction of the stent-graft delivery system.

Exclusion Criteria:

* Subject has a life expectancy < 2 years.
* Subject has a lesion that prevents safe delivery or expansion of the device.
* Subject has concomitant ascending aortic aneurysm.
* Subject has known allergies to any of the device materials.
* Subject has coagulopathy or bleeding disorders that cannot be pre-treated.
* Subject is contraindicated for contrast medium and anticoagulation drugs that cannot be pre-treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who experience ≥ 1 major adverse events (MAE) related to the experimental device/procedure at early (30-day) and late (6-month) endovascular TAA repair as compared with the open surgical repair group. | 30 day and 6 month
The primary effectiveness endpoint of early (30-day) and late (6-month) endovascular TAA repair will be assessed by the proportion of subjects free from major device related events | 30 day and 6 months

SECONDARY OUTCOMES:
• All cause mortality • Aneurysm related mortality compared to an open surgical control group • Major adverse events • Minor adverse events | 30 day and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Kartikeshwar Kasirajan, M.D., Principal Investigator — Emory University Medical School
Locations (2):
- United States (2):
  - Christiana Hospital, Newark, Delaware
  - Emory University School of Medicine, Atlanta, Georgia